CLINICAL TRIAL: NCT06000761
Title: Frequent Standardized Oral Care Using Human Milk to Prevent Oral Dysbiosis and Improve Health Outcomes in Premature Infants in the Neonatal Intensive Care Unit
Brief Title: Frequent Standardized Oral Care Using Human Milk in the Neonatal Intensive Care Unit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 202101340
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Ventilator Associated Pneumonia; Bronchopulmonary Dysplasia; Respiratory Disease
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Bronchopulmonary Dysplasia; Respiration Disorders

STUDY DESIGN:
Intervention Model Description: The proposed study will prospectively follow 168 VLBW infants and 168 mothers (dyad) for 4 weeks following birth. Infants will be randomized into 1 of 3 groups. Standardized oral care will be performed every 3-4 hours using human milk (Group 1), every 3-4 hours using sterile water (Group 2) or every 12 hours using sterile water (Group 3).
Who Masked: Outcomes Assessor
Masking Description: All de-identified saliva and breast milk samples will be conducted at a UF lab outside of Shands. ETT culture samples will also be de-identified before sending to Shands CoreLab. Investigators determining clinical outcomes will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Standardized oral care performed every 3-4 hours using human milk, donor or breast milk.
  Interventions: Procedure: Standardized oral Care
- Group 2 (Active Comparator): Standardized oral care performed every 3-4 hours using sterile water.
  Interventions: Procedure: Standardized oral Care
- Group 3 (Active Comparator): Standardized oral care performed every 12 hours using sterile water.
  Interventions: Procedure: Standardized oral Care

INTERVENTIONS:
Procedure: Standardized oral Care — One sponge-tipped swab, saturated with sterile water or human milk, will used clean the oral cavity with 15 seconds each area. Surfaces include all 4 quadrants of the gum surface and upper posterior part of the oropharynx. A second swab, with sterile water or milk will be used on the ventral and posterior surfaces of the tongue. A third swab, saturated with sterile water or human milk, will be used to clean the outer surface of any dwelling oral tubes (endotracheal tube, NAVA or feeding tube). Lips will be cleaned with a sterile gauze saturated with sterile water or human milk. Oral cavity will be suctioned as needed with an oral suction devise to remove secretions.

SUMMARY:
Premature infants are susceptible to complications related to infrequent and non-standardized oral care. Although the benefits of frequent standardized oral care are known to reduce oral dysbiosis (increased level of potentially pathogenic bacteria) and its associated complications in critically ill adults leading to established evidence-based guidelines, no such information exists for VLBW infants. The proposed study will prospectively follow 168 VLBW infants for 4 weeks following birth.

DETAILED DESCRIPTION:
Premature very low birth weight (VLBW) infants are susceptible to complications related to infrequent and non-standardized oral care. Although the benefits of frequent standardized oral care are known to reduce oral dysbiosis (increased level of potentially pathogenic bacteria) and its associated complications in critically ill adults leading to established evidence-based guidelines, no such information exists for VLBW infants. Premature VLBW infants are highly susceptible to costly, life threatening and potentially preventable morbidities, such as ventilator associated pneumonia (VAP), bronchopulmonary dysplasia (BPD; oxygen requirement at 28 days of life) and need for prolonged respiratory support which require additional treatments, increase cost of care, and can lead to chronic illness, re-hospitalization, and developmental delay. A dearth of information exists regarding oral care in VLBW infants, and no such guidelines exist for infants admitted to the neonatal intensive care unit (NICU) which may negatively affect their health. Thus, research regarding the effect of frequent, standardized oral care on the health of VLBW infants is essential to develop guidelines thus potentially improving the health of this vulnerable population. If successful, this research could change practice in NICUs across the nation.

ELIGIBILITY:
Inclusion:

* Mother ≥18 years of age
* ≤ 30 weeks gestation
* Born weighing ≤ 1500 grams

Exclusion:

* Congenital anomalies of the face, lungs, or gastrointestinal system
* Not expected to live > 7 days following delivery.

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 218 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with oral microbiome dysbiosis. | 0-28 days
  Oral samples will be obtained weekly and the microbiome analyzed using rRNA 16s sequencing

SECONDARY OUTCOMES:
Number of participants with ventilator associated pneumonia | 0-28 days
  Evidence of ventilator pneumonia will be assessed weekly over the first 4 weeks of life
Number of participants with bronchopulmonary dysplasia | 0-60 days
  Evidence of bronchopulmonary dysplasia will be assessed weekly over the first 60 days of life
Number of days requiring respiratory support | 0-60 days
  Days the infant was on any type of respiratory support will be assessed daily for the first 60 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Parker, PHD, Principal Investigator — University of Florida
Locations (1):
- Neonatal intensive care unit at Shands children's hospital at the Univeristy of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT06000761/Prot_000.pdf